CLINICAL TRIAL: NCT00903162
Title: Extended Endocrine Therapy for Premenopausal Women With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Ann H. Partridge, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-280
Record Dates: First submitted 2009-05-05; First posted 2009-05-18 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: hormone-receptor positive; tamoxifen; letrozole; zoledronic acid; leuprolide
MeSH Terms: conditions — Breast Neoplasms | interventions — Leuprolide; Letrozole; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Letrozole-Leuprolide (Experimental): Patients will receive 2.5mg oral letrozole daily and either 7.5mg monthly of Leuprolide IM or 22.5mg every three months of Leuprolide IM. Zoledronic acid 4mg IV every 6 months x 4 will also be offered optionally.
  Interventions: Drug: leuprolide; Drug: letrozole; Drug: zoledronic acid

INTERVENTIONS:
Drug: leuprolide — Given intramuscularly beginning on day 1 and then either 7.5 mg every month or 22.5 mg every 3 months for two years
  Other Names: Lupron
Drug: letrozole — Taken orally once a day 6-8 weeks after initial leuprolide administration
  Other Names: Femara
Drug: zoledronic acid — If desired, given intravenously every 6 months for a total of 4 injections (optional)
  Other Names: Zometa

SUMMARY:
The purpose of this study is to determine the safety and tolerability of the combination of two drugs (letrozole and leuprolide) in women who have already taken tamoxifen for at least 4.5 years. Letrozole, an aromatase inhibitor (which blocks an enzyme that produces estrogen), is a drug that is FDA approved. It has been shown to reduce the risk of breast cancer recurrence in postmenopausal women with breast cancer who have been previously treated with tamoxifen. Letrozole works by stopping the production of estrogen in parts of the body other than the ovaries. Leuprolide is a drug that stops a women's ovarian cycles. This process is known as ovarian function suppression. Stopping a women's menstrual cycle may be effective against breast cancer for some patients when given as initial therapy. The combination of letrozole and leuprolide is considered a standard treatment for women with metastatic breast cancer, and is also sometimes used for treatment of premenopausal early stage breast cancer, but it has not been accepted as a standard of care treatment.

DETAILED DESCRIPTION:
* Participants will be given a monthly intramuscular injection of leuprolide. Six to eight weeks after the first leuprolide injection, participants will be instructed to begin taking letrozole pills by mouth at home each day.
* During this research study, participants will also be offered injections of zoledronic acid to preserve bone mineral density. If desire, these injections will be given every 6 months for a total of 4 injections during the course of the research study.
* The treatments in this research study may increase the risk of bone density loss, so vitamin D and calcium supplements will be recommended to participants.
* The following tests and procedures will be performed during the research study: Physical Exam (every visit); Blood tests; Urine test (beginning and end of treatment); Imaging (annual mammograms); Bone Density (DXA) Scan (beginning and end of treatment); Questionnaires (throughout the study).
* Participants will be on this study for about two years.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older
* History of invasive ER+ or PR+ breast cancer treated with at least 4.5 years of tamoxifen
* No current evidence of recurrent invasive disease or metastatic disease. Patients may have a history of bilateral breast cancer
* Premenopausal (estradiol level in premenopausal range, >20pg/ml, within the prior 28 days)
* Liver function tests and creatinine <2.5 times the upper limit of normal within the 28 days prior to enrollment
* ECOG Performance Status 0-1
* Must agree to use non-hormonal contraception (condoms, diaphragm, IUD, sterilization, abstinence, etc) and no other hormonal therapy during trial and until 3 months after letrozole is stopped
* Negative pregnancy test within 14 days prior to enrollment
* Patient must be able to speak, read and write in English

Exclusion Criteria:

* Previous treatment with an oral or IV bisphosphonate in the prior two years
* History of cancer other than breast cancer within 5 years excluding basal/squamous cell skin carcinoma in situ of the cervix
* Women with evidence of current local recurrence or metastatic breast cancer
* Pregnant women
* Nursing women
* Women who are currently taking tamoxifen and are unwilling to stop this medication
* Women with a known deleterious BRCA 1 or BRCA 2 mutation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-05; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Partridge, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - University of Colorado, Denver, Colorado
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Newton Wellesley Hospital, Newton, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential patients were approached in the Dana-Farber Breast Oncology clinic and Newton Wellesley Hospital. Eligible patients were then presented with the study and given an opportunity to sign consent. The recruitment period ran from March 30th 2009 to May 1st, 2012.
Pre-assignment Details: A total of 17 patients were enrolled in this study; however, only 16 patients started treatment. One patient withdrew from the study before starting treatment.
Period: Overall Study
Arm/Group | Letrozole-Leuprolide
Started | 16
Completed | 12
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Enrolled participants.
Arm/Group | Letrozole-Leuprolide
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Tolerability at One Year of Ovarian Function Suppression (OFS) Using Leuprolide and Letrozole.
Description: The tolerability at one year of ovarian function suppression (OFS) using leuprolide and letrozole in this patient population. Specifically, the number of patients who discontinued treatment prior to one year due to toxicity.
Time Frame: 1 year
Population: Between September 15, 2009, and January 18, 2013, 17 patients were enrolled, but only 16 actually began protocol-directed treatment. Of the 16, 4 stopped treatment before completing even 1 year of protocol-directed therapy, owing to toxicity.
Measure: Number; unit: participants
Arm/Group | Letrozole-Leuprolide
Number analyzed (Participants) | 16
participants | 4

2. Secondary Outcome: Ovarian Function Suppression (OFS) Combined With Aromatase Inhibition Combined With Intravenous Bisphosphonate Therapy on Bone Mineral Density.
Description: Ovarian function suppression (OFS) combined with aromatase inhibition combined with intravenous bisphosphonate therapy on bone mineral density in this patient population.
Time Frame: 2 years
Population: This data was not collected nor analyzed because of too few participants to be meaningful.
Arm/Group | Letrozole-Leuprolide
Number analyzed (Participants) | 0

3. Secondary Outcome: The Effect of OFS Combined With Aromatase Inhibitor Therapy on the Incidence and Severity of Menopausal Symptoms, Sexual Dysfunction, Musculoskeletal Complaints, Other Side Effects and Overall Quality of Life.
Description: OFS combined with aromatase inhibitor therapy on the incidence and severity of menopausal symptoms, sexual dysfunction, musculoskeletal complaints, other side effects and overall quality of life in this population.
Time Frame: 2 years
Population: This data was not collected nor analyzed because of too few participants to be meaningful.
Arm/Group | Letrozole-Leuprolide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for the two years that patients were on study treatments.
Description: Adverse events data were collected from all participants enrolled in the study.
Arm/Group | Letrozole-Leuprolide
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 12/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole-Leuprolide (N=17)
Hot Flashes (Endocrine disorders) | 12 (12) — Hot Flashes/Flushes
Vaginal Dryness (Reproductive system and breast disorders) | 11 (11) — Dryness of the vagina
Headache (Nervous system disorders) | 6 (6) — disorder characterized by a sensation of marked discomfort in various parts of the head, not confined to the area of distribution of any nerve.
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (12) — Muscle pain
Flu-like Symptoms, Fever, or Rigors (General disorders) | 2 (2) — A disorder characterized by a group of symptoms similar to those observed in patients with the flu. It includes fever, chills, body aches, malaise, loss of appetite and dry cough.
Nausea (Gastrointestinal disorders) | 3 (3) — A disorder characterized by a queasy sensation and/or the urge to vomit.
Insomnia (Psychiatric disorders) | 3 (3) — A disorder characterized by difficulty in falling asleep and/or remaining asleep.
Fatigue (General disorders) | 6 (6) — A disorder characterized by a state of generalized weakness with a pronounced inability to summon sufficient energy to accomplish daily activities.
Sexual Dysfunction (Reproductive system and breast disorders) | 4 (4) — A disorder characterized by a decrease in sexual desire or function.
Injection Site Reaction or Rash (General disorders) | 3 (3) — A disorder characterized by an intense adverse reaction (usually immunologic) developing at the site of an injection.
Vaginal Discharge (Reproductive system and breast disorders) | 2 (2) — A disorder characterized by vaginal secretions. Mucus produced by the cervical glands is discharged from the vagina naturally, especially during the childbearing years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No